CLINICAL TRIAL: NCT04523714
Title: Tailored Non-Pharmacotherapy Services for Chronic Pain: Testing Scalable and Pragmatic Approaches
Brief Title: Tailored Non-Pharmacotherapy Services for Chronic Pain
Acronym: RESOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Essentia Health (Other); Georgia State University (Other); Duke University (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 192317
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: nonpharmacologic treatment; cognitive behavioral therapy; telehealth
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study uses a 3-arm, parallel intervention design; both intervention arms will be compared to usual care services.
Who Masked: Outcomes Assessor
Masking Description: Primary and secondary outcome assessors will be masked to treatment assignment. It is not feasible for participants to be masked to treatment arm assignment due to the type of intervention. The PI and select Co-Investigators and study staff who are involved in the oversight and delivery of the interventions will also be aware of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online CBT-CP based program (Active Comparator): Self-completed, online program in which participants complete eight, interactive sessions (approximately one per week) focused on training in one or more evidence-based pain coping skills (no usual care services restricted)
  Interventions: Behavioral: Online CBT-CP based program
- Virtual health coach-led CBT-CP based program (Active Comparator): Live, health coach-led program delivered by telephone or videoconference in which participants complete eight, interactive sessions (approximately one per week) focused on training in one or more evidence-based pain coping skills (no usual care services restricted)
  Interventions: Behavioral: Virtual health coach-led CBT-CP based program
- Usual Care plus information (No Intervention): Receipt of a bound copy of the 2020 edition of the American Chronic Pain Association Resource Guide to Chronic Pain Management and any pharmacologic and nonpharmacologic treatments available to them without restriction

INTERVENTIONS:
Behavioral: Online CBT-CP based program — Self-completed, online program in which participants complete eight, interactive sessions (approximately one per week) focused on training in one or more evidence-based pain coping skills
  Arms: Online CBT-CP based program
Behavioral: Virtual health coach-led CBT-CP based program — Live, health coach-led program delivered by telephone or videoconference in which participants complete eight, interactive sessions (approximately one per week) focused on training in one or more evidence-based pain coping skills
  Arms: Virtual health coach-led CBT-CP based program

SUMMARY:
The RESOLVE study is a multicenter comparative effectiveness trial of two cognitive behavioral therapy-based chronic pain (CBT-CP) treatments delivered via telehealth modalities: 1) online program and 2) live, health coach-led, virtual sessions (telephone and/or video conference).

DETAILED DESCRIPTION:
Specific Aims Aim #1: Determine the effectiveness of an online, CBT-based pain management program and virtual coach-led (telephonic/video) CBT-CP on achieving clinically meaningful improvements in patients' pain severity (pain intensity + pain-related interference) relative to those receiving usual care at 3 months.

1a. Examine the impact of the active interventions on secondary pain outcomes and related quality of life outcomes (social role functioning, physical functioning, and patient global impression of change); as well as exploratory outcomes, which include long-term opioid use; comorbid symptomology (depression, anxiety, and sleep disturbance); and high impact chronic pain and graded chronic pain.

1b. Conduct subgroup analyses to determine the impact of the active interventions on specific populations and explore for potential heterogeneity of treatment effects by sex; rural/medically underserved residency; multiple pain conditions; mental health mood disorders; and negative social determinants of health.

1c. Examine the role of theory-based mediators, pain catastrophizing, pain-related self-efficacy, and perceived support, on pain-severity.

Aim #2: Assess the cost and incremental cost-effectiveness of the online and virtual coach-led CBT-CP interventions compared to each other and usual care.

Aim #3: Conduct a qualitative evaluation to understand: 1) patient experiences of the interventions, including how they relate to treatment response, variability by site, and rural/medically underserved residency status; and 2) health system issues, including adaptations and contextual factors at the site and external levels, barriers and facilitators to intervention success and potential for adoption, sustainability and dissemination.

ELIGIBILITY:
INCLUSION CRITERIA

Electronic Health Record-based inclusion criteria:

* Active/enrolled in one of the 4 participating integrated health care systems at the time of query and for the prior 360 days
* Age 18 years or older (based on date of birth documented in EHR)
* English speaking or do not need interpreter services
* Have at least one [at Essentia] or at least two which are >60 days apart [at KP sites] outpatient pain-related health care encounter with nonmalignant musculoskeletal pain diagnoses [as determined by ICD10 codes for any of the following: back-neck-, limb/extremity-, joint-pain, arthritic disorders, fibromyalgia, headache, orofacial/temporomandibular pain, or musculoskeletal pain] within the past 360 days
* Do not have an encounter for surgery related to common musculoskeletal pain conditions (e.g., joint replacement, spinal fusion, carpal tunnel release surgery) [as determined by CPT and/or ICD-10 codes] within the past 60 days
* Do not have two or more separate encounters with a malignant cancer diagnosis other than non-melanoma skin cancer [as determined by ICD-10 codes] within past 60 days
* Do not have ICD-10 code(s), Current Procedural Terminology (CPT) code(s) or department/provider encounters indicating receipt of hospice or other palliative care within the past 360 days
* Do not have ICD-10 codes indicating severe cognitive impairment precluding participation in a behavioral/ lifestyle change program
* Note: At the KPWA site only, one additional EHR-based exclusion criterion will be applied, which is: Do not have ICD-10 codes indicating opioid use disorder (OUD). This criterion is being applied because there is another HEAL study being conducted at KPWA that focuses on treating individuals with pain and OUD specifically.]

Patient-reported inclusion criteria:

* Have high-impact chronic pain (as indicated by self-report of having pain on most or every day in past 3 months and pain limiting life or work activities on most or every day in past 3 months)
* Have persistent pain (as indicated by self-report Pain, Enjoyment of Life and General Activity (PEG) score of ≥ 12)
* Be able to participate in either of the active interventions (i.e., have internet and phone access required for accessing treatments)

EXCLUSION CRITERIA (patient-reported):

* Have received CBT for pain or pain-related psychoeducation or behavioral skills training within in the past 6 months (in-person, by phone or videoconference, or online)
* Currently receiving or will be starting CBT for pain or pain-related psychoeducation or behavioral skills training in the next month (in-person, by phone or videoconference, or online)
* Currently receiving or will be starting inpatient or intensive outpatient services for substance use disorder in the next month
* Have a planned/scheduled surgery in next 12 months related to pain condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2333 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn L DeBar, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (4):
- United States (4):
  - Kaiser Permanente Georgia, Center for Research and Evaluation, Atlanta, Georgia
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Kaiser Permanente Northwest Center for Health Research, Portland, Oregon
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
A releasable database containing underlying Individual Participant Data (IPD) from the primary outcomes manuscript and all National Institutes of Health (NIH) HEAL (Helping to End Addiction Long-term) Initiative common data elements will be produced and made broadly available through the NIH HEAL Initiative-designated central data repository. The database will be completely de-identified in accordance with the definitions provided in the Health Insurance Portability and Accountability Act (HIPAA) and in accordance to the standards set forth in the Department of Health and Human Services Regulations for the Protection of Human Subjects. Namely, all identifiers specified in HIPAA will be recoded in a manner that will make it impossible to deduce or impute the specific identity of any patient. The database will not contain any institutional or healthcare system identifiers.
Supporting Information: Study Protocol
Time Frame: The database will be released at the time of publication of the primary manuscript, or within 12 months of last patient procedure, whichever comes first. The duration of availability will be in accordance with procedures and regulations of the NIH HEAL Initiative and the project funder (NIA).
Access Criteria: Access to the releasable database housed in the NIH-assigned repository will be in accordance with procedures and regulations of the NIH HEAL Initiative and the project funder (NIA).

REFERENCES:
- [Background] DeBar LL, Mayhew M, Wellman RD, Balderson BH, Dickerson JF, Elder CR, Justice M, Keefe FJ, McMullen CK, Owen-Smith AA, Rini C, Von Korff M, Waring S, Yarava A, Shen Z, Thompson RE, Clark AE, Casper TC, Cook AJ. Telehealth and Online Cognitive Behavioral Therapy-Based Treatments for High-Impact Chronic Pain: A Randomized Clinical Trial. JAMA. 2025 Jul 23;334(7):592-605. doi: 10.1001/jama.2025.11178. Online ahead of print. PMID 40699570
- [Background] Mayhew M, Balderson BH, Cook AJ, Dickerson JF, Elder CR, Firemark AJ, Haller IV, Justice M, Keefe FJ, McMullen CK, O'Keeffe-Rosetti MC, Owen-Smith AA, Rini C, Schneider JL, Von Korff M, Wandner LD, DeBar LL. Comparing the clinical and cost-effectiveness of remote (telehealth and online) cognitive behavioral therapy-based treatments for high-impact chronic pain relative to usual care: study protocol for the RESOLVE multisite randomized control trial. Trials. 2023 Mar 16;24(1):196. doi: 10.1186/s13063-023-07165-8. PMID 36927459

RESULTS

PARTICIPANT FLOW:
Groups:
- Online CBT-CP Based Program: Self-completed, online cognitive behavioral therapy for chronic pain (CBT-CP)-based skills training program in which participants complete eight, interactive sessions (approximately one per week) focused on training in one or more evidence-based CBT-CP skills (no usual care services restricted)
- Health Coach-led CBT-CP Based Program: Live, coach-led cognitive behavioral therapy for chronic pain (CBT-CP)-based skills training program delivered by telephone or videoconference in which participants complete eight, interactive sessions (approximately one per week) focused on training in one or more evidence-based CBT-CP skills (no usual care services restricted)
Period: Overall Study
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Started | 776 | 778 | 779
Completed | 730 | 726 | 754
Not Completed | 46 | 52 | 25
Not completed — Death | 3 | 7 | 7
Not completed — Withdrawal by Subject | 43 | 45 | 16
Not completed — Randomized in error | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The 2 individuals randomized in error are not reported/included in the Baseline Analysis Population as they were not eligible (i.e., 779 in the Usual Care Plus in the Participant Flow vs. 777 in Baseline Analysis Population).
  The 2 individuals who were randomized in error (i.e., totaling 2,333 in the Participant Flow) were withdrawn immediately after randomization when the error was identified. That is why the Baseline Analytic Population = 2,331.
Groups:
- Total: Total of all reporting groups
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information | Total
Number analyzed (Participants) | 776 | 778 | 777 | 2331
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (13.9) | 58.8 (14.5) | 58.8 (14.3) | 58.8 (14.3)
Age, Customized [Count of Participants; unit: Participants]
  Age 65 years and older | 291 | 305 | 304 | 900
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 571 | 572 | 570 | 1713
  Male | 205 | 206 | 207 | 618
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity : White Non-Hispanic | 573 | 572 | 554 | 1699
  Race and Ethnicity : Black or African American Non-Hispanic | 119 | 118 | 113 | 350
  Race and Ethnicity : Hispanic | 21 | 26 | 30 | 77
  Race and Ethnicity : Asian | 10 | 6 | 11 | 27
  Race and Ethnicity : American Indian / Alaska Native | 6 | 11 | 11 | 28
  Race and Ethnicity : Native Hawaiian / Other Pacific Islander | 1 | 0 | 1 | 2
  Race and Ethnicity : More than one race | 21 | 27 | 35 | 83
  Missing | 25 | 18 | 22 | 65
Region of Enrollment [Number; unit: participants]
  United States | 776 | 778 | 777 | 2331
Rural/medically underserved residency [Count of Participants; unit: Participants] | 340 | 345 | 345 | 1030

OUTCOME MEASURES:

1. Primary Outcome: Minimal Clinically Important Difference (MCID) in Pain Severity at 3 Months (Yes / No)
Description: Minimal clinically important difference (MCID) in pain severity is defined as a 30% or greater improvement in pain severity score. [Pain severity score assessed via modified 11-item version of the Brief Pain Inventory - Short Form (BPI-SF) from baseline (consistent with IMMPACT guidelines). The BPI-SF range= 0 to 10; higher score = worse pain severity.]
  MCID outcome is binary; reported as the adjusted percentage of participants with MCID (> or =30% improvement) in pain severity.
Time Frame: Baseline to 3 months
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of participants
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 776 | 778 | 777
Adjusted percentage of participants | 26.6 [23.4 to 30.2] | 32.0 [29.3 to 35.0] | 20.8 [18.0 to 24.0]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment (see SAP); Relative Risk = 1.28, 95% CI 2-sided [1.06 to 1.55]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment; Relative Risk = 1.54, 95% CI 2-sided [1.30 to 1.82]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment (See SAP); Relative Risk = 1.20, 95% CI 2-sided [1.03 to 1.40]

2. Secondary Outcome: MCID in Pain Severity at 6 Months (Yes / No)
Description: Minimal clinically important difference (MCID) in pain severity is defined as a 30% decrease in score on modified 11-item version of the Brief Pain Inventory - Short Form (BPI-SF) from baseline (consistent with IMMPACT guidelines) (binary)
  Minimal clinically important difference (MCID) in pain severity is defined as a 30% or greater improvement in pain severity score. [Pain severity score assessed via modified 11-item version of the BPI-SF from baseline (consistent with IMMPACT guidelines). The BPI-SF range= 0 to 10; higher score = worse pain severity.]
  MCID outcome is binary; reported as the adjusted percentage of participants with MCID (> or =30% improvement) in pain severity.
Time Frame: Baseline to 6 months
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of participants
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 776 | 778 | 777
Adjusted percentage of participants | 32.9 [29.5 to 36.7] | 37.1 [34.1 to 40.5] | 22.9 [20.0 to 26.1]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment (see SAP); Relative Risk = 1.44, 95% CI 2-sided [1.21 to 1.70]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment (see SAP); Relative Risk = 1.62, 95% CI 2-sided [1.39 to 1.90]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment (see SAP); Relative Risk = 1.13, 95% CI 2-sided [0.98 to 1.30]

3. Secondary Outcome: MCID in Pain Severity at 12 Months (Yes / No)
Description: Minimal clinically important difference (MCID) in pain severity is defined as a 30% or greater improvement in pain severity score. [Pain severity score assessed via modified 11-item version of the BPI-SF from baseline (consistent with IMMPACT guidelines). The BPI-SF range= 0 to 10; higher score = worse pain severity.]
  MCID outcome is binary; reported as the adjusted percentage of participants with MCID (> or =30% improvement) in pain severity.
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of participants
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 776 | 778 | 777
Adjusted percentage of participants | 35.9 [32.4 to 39.7] | 38.3 [36.8 to 39.9] | 27.1 [24.1 to 30.5]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment (see SAP); Relative Risk = 1.32, 95% CI 2-sided [1.13 to 1.54]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment (see SAP); Relative Risk = 1.41, 95% CI 2-sided [1.25 to 1.59]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Test type: Superiority; p < 0.001, Modified Poisson Regression — A priori threshold for statistical significance <0.05; Imputation, weighting and adjustment; Relative Risk = 1.07, 95% CI 2-sided [0.96 to 1.19]

4. Secondary Outcome: Pain Severity Score
Description: Modified 11-item version of the Brief Pain Inventory - Short Form (BPI-SF). Score is calculated mean of all 11 items; range 0-10 with a higher score = worse pain severity
Time Frame: Baseline to 3, 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: Adjusted mean change (score on a scale)
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 643 | 690 | 703
Adjusted mean change (score on a scale)
  3 months | -1.2 [-1.3 to -1.0] | -1.2 [-1.3 to -1.1] | -0.8 [-0.9 to -0.6]
  6 months | -1.3 [-1.4 to -1.1] | -1.4 [-1.5 to -1.3] | -0.9 [-1.0 to -0.8]
  12 months | -1.5 [-1.6 to -1.3] | -1.4 [-1.6 to -1.3] | -1.1 [-1.2 to -0.9]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear; Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear; Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.3]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear; Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Median Difference (Final Values) = -0.0, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 4: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2]
Statistical Analysis 5: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.4]
Statistical Analysis 6: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 7: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2]
Statistical Analysis 8: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2]
Statistical Analysis 9: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

5. Secondary Outcome: Pain Intensity Score
Description: 4-item subscale of the Brief Pain Inventory - Short Form (BPI-SF). Score is calculated mean of all 4 items; range 0-10 with a higher score = worse pain intensity
Time Frame: Baseline to 3, 6, and 12 months
Measure: Mean (95% Confidence Interval); unit: Adjusted mean change (score on a scale)
Arm/Group | Online CBT-CP Based Program | Virtual Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 643 | 690 | 703
Adjusted mean change (score on a scale)
  3 months | -0.9 [-1.0 to -0.8] | -0.9 [-1.0 to -0.8] | -0.6 [-0.7 to -0.5]
  6 months | -1.0 [-1.1 to -0.9] | -1.1 [-1.2 to -1.0] | -0.7 [-0.9 to -0.6]
  12 months | -1.1 [-1.3 to -1.0] | -1.1 [-1.3 to -1.0] | -0.9 [-1.0 to -0.8]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear; Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.1]
Statistical Analysis 2: Comparison: Virtual Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.2]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Virtual Health Coach-led CBT-CP Based Program; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 4: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); p < 0.05, GEE, linear; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1]
Statistical Analysis 5: Comparison: Virtual Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.2]
Statistical Analysis 6: Comparison: Online CBT-CP Based Program vs Virtual Health Coach-led CBT-CP Based Program; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 7: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1]
Statistical Analysis 8: Comparison: Virtual Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); p < 0.05, GEE, linear; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1]
Statistical Analysis 9: Comparison: Online CBT-CP Based Program vs Virtual Health Coach-led CBT-CP Based Program; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

6. Secondary Outcome: Pain-related Interference Score
Description: 7-item subscale of the Brief Pain Inventory - Short Form (BPI-SF). Score is calculated mean of 7 items; range 0-10 with a higher score = worse pain-related interference
Time Frame: Baseline to 3, 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: Adjusted mean change (score on a scale)
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 643 | 690 | 703
Adjusted mean change (score on a scale)
  3 months | -1.3 [-1.4 to -1.1] | -1.4 [-1.5 to -1.2] | -0.8 [-1.0 to -0.7]
  6 months | -1.5 [-1.6 to -1.3] | -1.6 [-1.8 to -1.4] | -1.0 [-1.1 to -0.8]
  12 months | -1.6 [-1.8 to -1.5] | -1.6 [-1.8 to -1.5] | -1.2 [-1.3 to -1.0]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.3]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.3]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 4: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.3]
Statistical Analysis 5: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.8 to -0.4]
Statistical Analysis 6: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 7: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.3]
Statistical Analysis 8: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.3]
Statistical Analysis 9: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

7. Secondary Outcome: Social Role Functioning
Description: PROMIS Ability to Participate in Social Roles and Activities - Short Form 4a: Score by summing the 4 items (each item response 1-5) and then converting raw score to standardized T-score, using the HealthMeasures Scoring Service, with mean of 50 and standard deviation of 10. Higher T-score= better ability to participate in social roles and activities. Score ≤40 indicates moderate (40-30) to severe (< 30) limitations in ability to participate.
Time Frame: Baseline to 3, 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: Adjusted mean change (score on a scale)
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 636 | 683 | 696
Adjusted mean change (score on a scale)
  3 months | 1.5 [1.0 to 2.1] | 2.2 [1.7 to 2.7] | 0.7 [0.3 to 1.2]
  6 months | 2.2 [1.6 to 2.8] | 2.5 [2.0 to 3.1] | 1.0 [0.5 to 1.5]
  12 months | 2.6 [2.0 to 3.2] | 2.7 [2.2 to 3.3] | 1.4 [0.8 to 1.9]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.0 to 1.5]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 1.5, 95% CI 2-sided [0.8 to 2.2]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.7, 95% CI 2-sided [0.0 to 1.4]
Statistical Analysis 4: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.4 to 1.9]
Statistical Analysis 5: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 1.5, 95% CI 2-sided [0.8 to 2.2]
Statistical Analysis 6: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.4 to 1.1]
Statistical Analysis 7: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.5 to 2.1]
Statistical Analysis 8: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.6 to 2.1]
Statistical Analysis 9: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.7 to 0.9]

8. Secondary Outcome: Physical Functioning
Description: PROMIS Physical Function - Short Form 6b: Score by summing the 6 items (each item response 1-5) and then converting raw score to standardized T-score, using the HealthMeasures Scoring Service, with mean of 50 and standard deviation of 10. Higher T-score= better physical functioning. Score ≤40 indicates moderate (40-30) to severe (< 30) limitations in physical functioning.
Time Frame: Baseline to 3, 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: Adjusted mean change (score on a scale)
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 639 | 684 | 699
Adjusted mean change (score on a scale)
  3 months | 1.4 [1.1 to 1.8] | 1.7 [1.4 to 2.1] | 1.0 [0.7 to 1.4]
  6 months | 2.0 [1.6 to 2.4] | 1.8 [1.4 to 2.1] | 1.4 [1.0 to 1.7]
  12 months | 2.2 [1.8 to 2.7] | 2.1 [1.7 to 2.5] | 1.3 [0.9 to 1.7]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equation (GEE); Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.7, 95% CI 2-sided [0.2 to 1.2]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equation (GEE); Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 4: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equation (GEE); Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.1 to 1.2]
Statistical Analysis 5: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equation (GEE); Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 6: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equation (GEE); Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 7: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equation (GEE); Mean Difference (Final Values) = 0.9, 95% CI 2-sided [0.3 to 1.5]
Statistical Analysis 8: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equation (GEE); Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.2 to 1.4]
Statistical Analysis 9: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equation (GEE); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.5]

9. Secondary Outcome: Patient Global Impression of Change (PGIC) - Pain
Description: One item assessing participant's perception of change in pain since start of study; range 1-7 (1=much better, 2=moderately better, 3=a little better, 4=No change, 5=a little worse, 6=moderately worse, 7=much worse). Higher score = worsening of pain
Time Frame: Primary: Baseline to 3, 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: Adjusted mean (score on a scale)
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 640 | 687 | 702
Adjusted mean (score on a scale)
  3 months | 2.2 [2.1 to 2.3] | 2.0 [1.9 to 2.1] | 2.9 [2.8 to 3.0]
  6 months | 2.2 [2.1 to 2.3] | 2.1 [2.0 to 2.2] | 2.8 [2.7 to 2.9]
  12 months | 2.2 [2.1 to 2.3] | 2.2 [2.1 to 2.4] | 2.8 [2.7 to 2.9]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-0.8 to -0.6]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.0 to -0.8]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.3 to -0.1]
Statistical Analysis 4: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.8 to -0.5]
Statistical Analysis 5: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-0.8 to -0.5]
Statistical Analysis 6: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 7: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.8 to -0.5]
Statistical Analysis 8: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.7 to -0.4]
Statistical Analysis 9: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.2]

10. Secondary Outcome: Patient Global Impression of Change (PGIC) - General
Description: One item assessing participant's perception of change in overall status since start of study; range 1-7 (1=much better, 2=moderately better, 3=a little better, 4=No change, 5=a little worse, 6=moderately worse, 7=much worse). Higher score = worsening of overall status
Time Frame: Baseline to 3, 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: Adjusted mean (score on a scale)
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
Number analyzed (Participants) | 640 | 687 | 702
Adjusted mean (score on a scale)
  3 months | 2.0 [1.9 to 2.1] | 1.6 [1.5 to 1.7] | 2.7 [2.6 to 2.8]
  6 months | 2.1 [2.0 to 2.2] | 1.8 [1.7 to 1.9] | 2.5 [2.5 to 2.6]
  12 months | 2.0 [1.9 to 2.1] | 1.9 [1.8 to 2.0] | 2.6 [2.5 to 2.7]
Statistical Analysis 1: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-0.8 to -0.6]
Statistical Analysis 2: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.2 to -1.0]
Statistical Analysis 3: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 3 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.5 to -0.3]
Statistical Analysis 4: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.6 to -0.3]
Statistical Analysis 5: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-0.9 to -0.6]
Statistical Analysis 6: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 6 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1]
Statistical Analysis 7: Comparison: Online CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.7 to -0.4]
Statistical Analysis 8: Comparison: Health Coach-led CBT-CP Based Program vs Usual Care Plus Information; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-0.8 to -0.5]
Statistical Analysis 9: Comparison: Online CBT-CP Based Program vs Health Coach-led CBT-CP Based Program; Baseline to 12 months; Test type: Superiority; p < 0.05, GEE, linear — Imputation, weighting and adjustment (see SAP). Generalized estimating equations (GEE); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0]

ADVERSE EVENTS:
Time Frame: 12-month study participation period
Description: Severe Adverse Events, including death and hospitalizations, were systematically monitored.
  Other Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
  These events were monitored for the 2,331 eligible randomized participants. The 2 individuals who were randomized in error (i.e., totaling 2,333 in the Participant Flow) were not monitored for these events as they were withdrawn immediately after randomization when the error was identified.
Arm/Group | Online CBT-CP Based Program | Health Coach-led CBT-CP Based Program | Usual Care Plus Information
All-Cause Mortality (participants affected / at risk) | 3/776 | 7/778 | 7/777
Serious Adverse Events (participants affected / at risk) | 55/776 | 65/778 | 63/777
Other Adverse Events (participants affected / at risk) | 1/776 | 16/778 | 0/777
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Online CBT-CP Based Program (N=776) | Health Coach-led CBT-CP Based Program (N=778) | Usual Care Plus Information (N=777)
Hospitalizations (General disorders) | 55 (81) | 65 (84) | 63 (82)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Online CBT-CP Based Program (N=776) | Health Coach-led CBT-CP Based Program (N=778) | Usual Care Plus Information (N=777)
Participant-reported adverse event (General disorders) | 1 (1) | 16 (16) | 0 (0) — Non-serious adverse events (AEs) were not systematically collected and only ascertained via patient-initiated report, biasing collection to the intervention groups which had more staff contact.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT04523714/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT04523714/SAP_001.pdf